CLINICAL TRIAL: NCT05308654
Title: First-in-Human Study of the BCL-2 Inhibitor ABBV-453 in Biomarker-Selected Subjects With Relapsed or Refractory Multiple Myeloma
Brief Title: A Study to Assess the Adverse Events and Change in Disease Activity in Adult Participants With Relapsed or Refractory Multiple Myeloma Receiving Oral ABBV-453 Tablets
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M21-406; 2022-501685-22 (Other: EU CT)
Record Dates: First submitted 2022-03-25; First posted 2022-04-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; ABBV-453; Cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Dexamethasone; daratumumab; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1: Monotherapy Dose Escalation (Experimental): Participants with relapsed or refractory (R/R) multiple myeloma (MM) will receive escalating doses of ABBV-453, until the maximum tolerated dose (MTD) is determined.
  Interventions: Drug: ABBV-453
- Part 2: Arm 1 (Experimental): Participants will receive continuous doses of ABBV-453 in combination with dexamethasone in 28-day cycles.
  Interventions: Drug: ABBV-453; Drug: Dexamethasone
- Part 2: Arm 2 (Experimental): Participants will receive continuous doses of ABBV-453 in combination with daratumumab and dexamethasone in 28-day cycles.
  Interventions: Drug: ABBV-453; Drug: Dexamethasone; Drug: Daratumumab
- Part 2: Arm 3 (Experimental): Participants will receive continuous doses of ABBV-453 in combination with daratumumab, lenalidomide, and dexamethasone in 28-day cycles.
  Interventions: Drug: ABBV-453; Drug: Dexamethasone; Drug: Daratumumab; Drug: Lenalidomide
- Japan Cohort (Experimental): Participants with R/R MM will receive escalating doses of ABBV-453, until the MTD is determined.
  Interventions: Drug: ABBV-453

INTERVENTIONS:
Drug: ABBV-453 — Oral; Tablet
Drug: Dexamethasone — Oral Tablet
  Arms: Part 2: Arm 1; Part 2: Arm 2; Part 2: Arm 3
Drug: Daratumumab — Subcutaneous Injection
  Arms: Part 2: Arm 2; Part 2: Arm 3
Drug: Lenalidomide — Oral Capsule
  Arms: Part 2: Arm 3

SUMMARY:
Multiple myeloma (MM) is a plasma cell disease characterized by the growth of clonal plasma cells in the bone marrow. The purpose of this study is to assess the safety and toxicity of ABBV-453 in adult participants with relapsed/refractory (R/R) MM. Adverse events and change in disease activity will be assessed.

ABBV-453 is an investigational drug being developed for the treatment of R/R MM. Part 1 will be a monotherapy dose escalation phase to determine the best dose of ABBV-453. In Part 2, participants are placed in 1 of 3 groups called treatment arms. Each group receives a different treatment. Approximately 28 to 48 adult participants in Part 1 and 150 to 312 adult participants in Part 2 with R/R MM will be enrolled in the study in approximately 70 sites worldwide.

In Part 1 and the Japan Cohort, Participants will receive oral ABBV-453 tablets once daily (QD) in 28-day cycles. In Part 2, Arm 1, participants will receive continuous doses of oral ABBV-453 tablets QD in combination with oral dexamethasone tablets once weekly in 28-day cycles. In Part 2, Arm 2, participants will receive continuous doses of oral ABBV-453 tablets QD in combination with subcutaneous injections of daratumumab every 1 to 4 weeks and oral dexamethasone tablets once weekly in, 28-day cycles. In Part 2, Arm 3, participants will receive continuous doses of oral ABBV-453 tablets QD in combination with subcutaneous injections of daratumumab every 1 to 4 weeks, oral lenalidomide capsules QD on Days 1-21, and oral dexamethasone tablets once weekly, in 28-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status <= 1.
* Laboratory values meeting the criteria outlined in the protocol.
* Documented diagnosis of multiple myeloma (MM) based on standard International Myeloma Working Group (IMWG) criteria.
* Has measurable disease at screening as defined in the protocol.
* Locally documented or centrally determined t(11;14) positive status and/or centrally determined BCL2high status. Note: If local testing for t(11;14) is discordant with central testing for t(11;14) status, a detailed review of central and local results for t(11;14) status is required to ensure the participants' safety.
* Part 1 and Part 2, Arm 1 Only: Refractory to or intolerant of all established MM therapies that are known to provide clinical benefit and are triple class exposed to a proteasome inhibitors (PI), an Immunomodulatory drugs (IMID), and an anti-CD38 monoclonal antibody in previous line(s) of therapy.
* Part 2, Arms 2 and 3 Only: Received 1 to 3 prior lines of therapy, including a PI or an IMiD.
* Part 1 only: Permitted to be venetoclax or BCL-2 inhibitor exposed in previous lines of therapy.
* Life expectancy >= 12 weeks.

Exclusion Criteria:

* Clinically relevant or significant Electrocardiogram (ECG) abnormalities as outlined in the protocol.
* Part 2 only: Previous treatment with venetoclax or BCL-2 inhibitor.
* Part 2, Arms 2 and 3 only: Prior daratumumab or other anti-CD38 therapy exposure that meets any of the criteria outlined in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2024-02-07 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) per International Myeloma Working Group (IMWG) Criteria | Up to Approximately 12 Months
  ORR is defined as the percentage of participants with a confirmed best overall response (BOR) of partial response (PR) + very good partial response (VGPR) + complete response (CR) + stringent complete response (sCR) as assessed by investigators per adapted IMWG criteria for relapsed or refractory (R/R) multiple myeloma (MM).

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to Approximately 24 Months
  DOR is defined for participants achieving a confirmed sCR/CR/VGPR/PR as the time from the initial response of sCR/CR/VGPR/PR per investigator review according to adapted IMWG criteria to disease progression or death of any cause, whichever occurs earlier.
Depth of Response Minimal Residual Disease (MRD) | Up to Approximately 24 Months
  MRD negativity is defined as having less than 1 myeloma cell that may remain in the bone marrow aspirate. Depth of response is defined as the proportion of MRD negativity for participants achieving a confirmed sCR/CR per investigator review according to IMWG criteria.
Progression Free Survival (PFS) | Up to Approximately 36 Months
  PFS is defined as time from first study treatment to a documented disease progression according to adapted IMWG criteria, as determined by the investigator, or death due to any cause, whichever occurs earlier.
Overall Survival (OS) | Up to Approximately 36 Months
  Overall survival (OS) is defined as time from first study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (21):
- United States (12):
  - Stanford University School of Med /ID# 242809, Stanford, California
  - Sylvester Comprehensive Cancer Center /ID# 243417, Miami, Florida
  - Tulane University School of Medicine /ID# 244854, New Orleans, Louisiana
  - American Oncology Partners of Maryland /ID# 244858, Bethesda, Maryland
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 242754, Ann Arbor, Michigan
  - Mayo Clinic - Rochester /ID# 242844, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center /ID# 243503, New York, New York
  - Atrium Health Levine Cancer Institute /ID# 243420, Charlotte, North Carolina
  - Duke Univ Med Ctr /ID# 242808, Durham, North Carolina
  - Wake Forest Baptist Health /ID# 244252, Winston-Salem, North Carolina
  - University of Pennsylvania /ID# 242842, Philadelphia, Pennsylvania
  - Vanderbilt Ingram Cancer Center /ID# 242810, Nashville, Tennessee
- Australia (5):
  - Liverpool Hospital /ID# 244826, Liverpool, New South Wales
  - St. Vincent's Private Hospital Melbourne /ID# 262631, Fitzroy, Victoria
  - St Vincent's Hospital Melbourne /ID# 244827, Fitzroy Melbourne, Victoria
  - Austin Health and Ludwig Institute for Cancer Research /ID# 248311, Heidelberg, Victoria
  - Epworth Healthcare /ID# 248705, Richmond, Victoria
- Israel (3):
  - Hadassah Medical Center-Hebrew University /ID# 250484, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 250482, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 250483, Tel Aviv, Tel Aviv
- Barts Health NHS Trust /ID# 248972, London, London, City of, United Kingdom

IPD SHARING:
Plan to Share IPD: No